CLINICAL TRIAL: NCT02555683
Title: A 52-week, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of QAW039 When Added to Existing Asthma Therapy in Patients With Uncontrolled Severe Asthma.
Brief Title: Study of Efficacy and Safety of QAW039 in Patients With Severe Asthma Inadequately Controlled With Standard of Care Asthma Treatment.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAW039A2307; 2015-002553-35 (EudraCT Number)
Record Dates: First submitted 2015-09-18; First posted 2015-09-21 (Estimated); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-04

CONDITIONS: Asthma
Keywords: Asthma; QAW039; allergic asthma; allergy triggered asthma; reactive asthma; asthma attack; difficulty breathing
MeSH Terms: conditions — Asthma; Dyspnea | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- QAW039 150 mg (Experimental): QAW039 150 mg once daily
  Interventions: Drug: QAW039
- QAW039 450 mg (Experimental): QAW039 450 mg once daily
  Interventions: Drug: QAW039
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAW039 — QAW039 150 mg once daily
  Arms: QAW039 150 mg
Drug: QAW039 — QAW039 450 mg once daily
  Arms: QAW039 450 mg
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
This study aimed to determine the efficacy and safety of QAW039 150 mg and QAW039 450 mg, compared with placebo, when added to GINA (Global Initiative for Asthma) steps 4 and 5 standard-of- care (SoC) asthma therapy (GINA 2016) in the following two populations:

* patient with inadequately controlled severe asthma and high eosinophil counts at baseline (eosinophil count at Visit 1 ≥250 cells/ µl) (sub-population)
* patients with inadequately controlled severe asthma (overall study population)

Inadequate control is defined as partly controlled or uncontrolled asthma (GINA 2016).

DETAILED DESCRIPTION:
This study used a randomized, multicenter, double-blind, placebo-controlled parallel-group design in which QAW039 150 mg or QA039 450 mg or placebo was added to standard of care, GINA steps 4 and 5 asthma therapy.

The study included:

* Screening period of up to 2 weeks to assess eligibility;
* Run-in period of approximately 2 weeks and a maximum of 6 weeks on placebo to collect baseline data for efficacy variables and compliance with the Electronic Peak Flow/ eDiary device. Upon completion of the run-in period, all patients who met the eligibility criteria were randomized to one of three treatments: QAW039 150 mg or QAW039 450 mg or placebo once daily in a ratio of 1:1:1.
* Treatment period of 52 weeks (assessment period for all Primary and Secondary Outcome Measures). Clinic visits were scheduled approximately 4 weeks after randomization and then at approximately 8-week intervals during the active-treatment period. Phone calls occurred at specified time points between visits occurring at 8-week intervals. Patients who had successfully completed 52 weeks of treatment in this study were offered an optional participation in a safety study (CQAW039A2315).
* Follow-up period of 4 weeks, investigational and drug-free, following the last dose of study drug. A follow-up visit occurred approximately 4 weeks (i.e., approximately 30 days) following the last dose of study therapy to complete safety assessments and pregnancy testing (if applicable). the follow-up period applied to all patients except those patients who had entered the safety study (CQAW039A2315) directly after the Week 52 study visit.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and assent (if applicable).
* Male and female patients aged ≥12 years (or ≥lower age limit allowed by health authority and/or ethics committee/institutional review board approvals).
* A diagnosis of severe asthma, uncontrolled on GINA 4/5 asthma medication.
* Evidence of airway reversibility or airway hyper- reactivity.
* FEV1 of ≤80% of the predicted normal value for patients aged ≥18 years; FEV1 of ≤90% for patients aged 12 to <18 years
* An ACQ score ≥1.5.
* A history of 2 or more asthma exacerbations within the 12 months prior to entering the study.

Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives of study entry, or within 30 days, whichever is longer.
* Subjects who have participated in another trial of QAW039.
* A QTcF (Fridericia) ≥450 msec (male) or ≥460 msec (female).
* History of malignancy with the exception of local basal cell carcinoma of the skin.
* Pregnant or nursing (lactating) women.
* Serious co-morbidities.
* Patients on greater than 20 mg of simvastatin, greater than 40 mg of atorvastatin, greater than 40 mg of pravastatin, or greater than 2 mg of pitavastatin

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 894 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis
Locations (197):
- United States (52):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Gilbert, Arizona
  - Novartis Investigative Site, Litchfield Park, Arizona
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Hawaiian Gardens, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Redondo Beach, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Westminster, California
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Brandon, Florida
  - Novartis Investigative Site, New Smyrna Beach, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Ormond Beach, Florida
  - Novartis Investigative Site, Sebring, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Gainesville, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Crowley, Louisiana
  - Novartis Investigative Site, Zachary, Louisiana
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Gaithersburg, Maryland
  - Novartis Investigative Site, White Marsh, Maryland
  - Novartis Investigative Site, Livonia, Michigan
  - Novartis Investigative Site, Ypsilanti, Michigan
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, Bellevue, Nebraska
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Corning, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Gastonia, North Carolina
  - Novartis Investigative Site, Monroe, North Carolina
  - Novartis Investigative Site, New Bern, North Carolina
  - Novartis Investigative Site, Whiteville, North Carolina
  - Novartis Investigative Site, Wilmington, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Maumee, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Jefferson Hills, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, East Providence, Rhode Island
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Fairfax, Virginia
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As
- Australia (5):
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Footscray, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
- Austria (6):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Amstetten
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Thalheim bei Wels
  - Novartis Investigative Site, Vienna
- Belgium (9):
  - Novartis Investigative Site, Genk, Limburg
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Éghezée
  - Novartis Investigative Site, Herentals
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Ottignies
- Brazil (7):
  - Novartis Investigative Site, Porto Alegre, Porto Alegre RS
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, São Bernardo do Campo, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- China (16):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Haikou, Hainan
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chengdu
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Novartis Investigative Site, Copenhagen NV, Denmark
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (4):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, HUS
  - Novartis Investigative Site, OYS
  - Novartis Investigative Site, Tampere
- France (9):
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Strasbourg
- Germany (15):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Landsberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Neu-Isenburg
  - Novartis Investigative Site, Rosenheim
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Witten
- Novartis Investigative Site, Thessaloniki, GR, Greece
- Guatemala (3):
  - Novartis Investigative Site, Ciudad, Gautemala
  - Novartis Investigative Site, Guatemala City, GTM
  - Novartis Investigative Site, Guatemala City
- Hungary (8):
  - Novartis Investigative Site, Eger, HUN
  - Novartis Investigative Site, Győr, HUN
  - Novartis Investigative Site, Hajdúnánás, HUN
  - Novartis Investigative Site, Makó, HUN
  - Novartis Investigative Site, Százhalombatta, HUN
  - Novartis Investigative Site, Törökbálint, Pest County
  - Novartis Investigative Site, Komárom
  - Novartis Investigative Site, Pécs
- Novartis Investigative Site, Reykjavik, Iceland
- Novartis Investigative Site, Dublin, Ireland
- Latvia (2):
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Lithuania (6):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Klaipėda, LTU
  - Novartis Investigative Site, Vilnius, LTU
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
- Philippines (3):
  - Novartis Investigative Site, Bulacan
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Poland (5):
  - Novartis Investigative Site, Biaystok, Poland
  - Novartis Investigative Site, Kielce, POL
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Strzelce Opolskie
- Romania (11):
  - Novartis Investigative Site, Ploieşti, Prahova
  - Novartis Investigative Site, Constanța, ROM
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Arad
  - Novartis Investigative Site, Bragadiru
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Deva
  - Novartis Investigative Site, Oradea
  - Novartis Investigative Site, Sangiorgiu de Mures
- Singapore (2):
  - Novartis Investigative Site, Singapore, SGP
  - Novartis Investigative Site, Singapore
- Novartis Investigative Site, Barcelona, Spain
- Switzerland (5):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Liestal
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- United Kingdom (15):
  - Novartis Investigative Site, Cambridge, Cambrigdeshire
  - Novartis Investigative Site, Darlington, Durham
  - Novartis Investigative Site, London, GBR
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Chertsey
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Tyne and Wear
  - Novartis Investigative Site, Wakefield
  - Novartis Investigative Site, Wishaw
- Vietnam (3):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

REFERENCES:
- [Derived] Brightling CE, Gaga M, Inoue H, Li J, Maspero J, Wenzel S, Maitra S, Lawrence D, Brockhaus F, Lehmann T, Brindicci C, Knorr B, Bleecker ER. Effectiveness of fevipiprant in reducing exacerbations in patients with severe asthma (LUSTER-1 and LUSTER-2): two phase 3 randomised controlled trials. Lancet Respir Med. 2021 Jan;9(1):43-56. doi: 10.1016/S2213-2600(20)30412-4. Epub 2020 Sep 24. PMID 32979986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were from Argentina, Australia, Austria, Belgium, Brazil, China, Denmark, Estonia, Finland, France, Germany, Greece, Guatemala, Hungary, Latvia, Lithuania, Philippines, Poland, Romania, Singapore, Spain, Switzerland, UK, US, Vietnam.
Pre-assignment Details: The study included a Screening period of up to 2 weeks and a Placebo Run-in period of 2 to 6 weeks, during which eligibility for randomization was determined.
Period: Overall Study
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Started | 301 | 295 | 298
FAS/SAF: High Eosinophil Subpopulation (Full analysis set/safety set. All patients who received study drug and had high eosinophils count) | 200 | 201 | 201
FAS/SAF: Overall Population (Full analysis set/safety set. All patients who received study drug) | 299 | 293 | 298
Completed | 282 | 278 | 269
Not Completed | 19 | 17 | 29
Not completed — Physician Decision | 1 | 0 | 2
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Technical Problems | 1 | 1 | 0
Not completed — Protocol deviation | 0 | 1 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Death | 0 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Subject/guardian decision | 12 | 12 | 22
Not completed — Death post Treatment/safety period | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo | Total
Number analyzed (Participants) | 301 | 295 | 298 | 894
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (14.97) | 51.1 (14.29) | 50.3 (14.48) | 50.4 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 214 | 177 | 583
  Male | 109 | 81 | 121 | 311
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 214 | 215 | 213 | 642
  Black | 11 | 6 | 12 | 29
  Asian | 45 | 38 | 44 | 127
  Native American | 24 | 29 | 24 | 77
  Unknown | 1 | 2 | 3 | 6
  Other | 6 | 5 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Rate of Moderate-to-severe Asthma Exacerbations During the 52-week Treatment Period in High Eosinophils Subpopulation
Description: A severe asthma exacerbation is defined as treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days and hospitalization; or treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days and emergency department visit (greater than 24 hours*); or death due to asthma. A moderate asthma exacerbation is defined as treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days either as an outpatient or in emergency department visits (Emergency department visit less than or equal to 24 hours). The high eosinophils subpopulation consists of all patients with blood eosinophil count ≥ 250 cells/μL at baseline.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS) in high eosinophils subpopulation (count ≥ 250 cells/μL)
Measure: Least Squares Mean (95% Confidence Interval); unit: events/year
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 200 | 201 | 201
events/year | 0.97 [0.78 to 1.20] | 0.77 [0.62 to 0.97] | 0.93 [0.75 to 1.16]
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.800, negative binomial regression model — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; rate ratio = 1.04, 95% CI 2-sided [0.77 to 1.41]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.510, negative binomial regression model — adjusted p-value; Adjusted p-values are based on the closed testing procedure; Rate Ratio = 0.83, 95% CI 2-sided [0.61 to 1.14]

2. Secondary Outcome: Change From Baseline to Week 52 in Asthma Quality of Life Questionnaire for Participants 12 Years and Older (AQLQ+12) Score in High Eosinophils Subpopulation
Description: The AQLQ+12 is comprised of a total of 32 individual questions that span a total of four domains: symptoms, activity limitation, emotional function, and environmental stimuli.
  Patients were asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale (7 = not at all impaired to 1 = severely impaired). The AQLQ+12 yields individual domain scores, which is the mean of all items in each domain, and an overall score, which is the mean of all 32 individual responses. Higher scores indicate less impairment in health-related quality of life. The high eosinophils subpopulation consists of all patients with blood eosinophil count ≥ 250 cells/μL at baseline.
Time Frame: 52 weeks
Population: Full Analysis Set (FAS) in high eosinophils subpopulation (count ≥ 250 cells/μL)
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 200 | 201 | 201
units on scale | 0.75 (0.067) | 0.81 (0.067) | 0.68 (0.067)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.819, ANCOVA — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.11 to 0.26], Standard Error of Mean 0.095
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.591, ANCOVA — adjusted p-vale; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.05 to 0.32], Standard Error of Mean 0.095

3. Secondary Outcome: Change From Baseline to Week 52 in Asthma Control Questionnaire-5(ACQ-5) Score in High Eosinophils Subpopulation
Description: The ACQ-5 is a five-item, self-completed questionnaire, which is used as a measure of asthma control of a participant. Patients were asked to recall how their asthma had been during the previous week and to respond to the symptom questions on a 7-point scale (0=no impairment, 6=maximum impairment). The questions are equally weighted and the ACQ-5 score is the mean of the 5 questions: therefore, between 0 (totally controlled) and 6 (severely uncontrolled). The high eosinophils subpopulation consists of all patients with blood eosinophil count ≥ 250 cells/μL at baseline.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS) in high eosinophils subpopulation (count ≥ 250 cells/μL)
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 200 | 201 | 201
units on scale | -0.88 (0.069) | -0.94 (0.069) | -0.76 (0.070)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.819, ANCOVA — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.31 to 0.07], Standard Error of Mean 0.098
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.591, ANCOVA — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.37 to 0.02], Standard Error of Mean 0.098

4. Secondary Outcome: Change From Baseline to Week 52 in Pre-dose Forced Expiratory Volume in 1 Second (FEV1) in High Eosinophils Subpopulation
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline is defined as the last available FEV1 measurement taken prior to the first dose of randomized study drug. The high eosinophils subpopulation consists of all patients with blood eosinophil count ≥ 250 cells/μL at baseline.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS) in high eosinophils subpopulation (count ≥ 250 cells/μL)
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 200 | 201 | 201
Liter | 0.169 (0.0257) | 0.153 (0.0255) | 0.103 (0.0260)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.800, ANCOVA — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = 0.067, 95% CI 2-sided [-0.005 to 0.139], Standard Error of Mean 0.0365
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.523, ANCOVA — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = 0.050, 95% CI 2-sided [-0.021 to 0.121], Standard Error of Mean 0.0363

5. Primary Outcome: Rate of Moderate-to-severe Asthma Exacerbations During the 52-week Treatment Period in Overall Population
Description: A severe asthma exacerbation is defined as treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days and hospitalization; or treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days and emergency department visit (greater than 24 hours*); or death due to asthma. A moderate asthma exacerbation is defined as treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days either as an outpatient or in emergency department visits (Emergency department visit less than or equal to 24 hours).
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS) in overall population
Measure: Least Squares Mean (95% Confidence Interval); unit: events/year
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 299 | 293 | 298
events/year | 0.92 [0.77 to 1.09] | 0.75 [0.62 to 0.90] | 0.96 [0.80 to 1.15]
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.819, negative binomial regression model — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; rate ratio = 0.96, 95% CI 2-sided [0.75 to 1.22]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.510, negative binomial regression model — adjusted p-value; Adjusted p-values are based on the closed testing procedure; Rate Ratio = 0.78, 95% CI 2-sided [0.61 to 1.01]

6. Secondary Outcome: Change From Baseline to Week 52 in Asthma Quality of Life Questionnaire for Participants 12 Years and Older (AQLQ+12) Score in Overall Population
Description: The AQLQ+12 is comprised of a total of 32 individual questions that span a total of four domains: symptoms, activity limitation, emotional function, and environmental stimuli.
  Patients were asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale (7 = not at all impaired to 1 = severely impaired). The AQLQ+12 yields individual domain scores, which is the mean of all items in each domain, and an overall score, which is the mean of all 32 individual responses. Higher scores indicate less impairment in health-related quality of life.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS) in overall population
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 299 | 293 | 298
units on scale | 0.68 (0.053) | 0.73 (0.054) | 0.61 (0.054)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.819, ANCOVA — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.07 to 0.23], Standard Error of Mean 0.076
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.591, ANCOVA — adjusted p-vale; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.03 to 0.27], Standard Error of Mean 0.076

7. Secondary Outcome: Change From Baseline to Week 52 in Asthma Control Questionnaire-5(ACQ-5) Score in Overall Population
Description: The ACQ-5 is a five-item, self-completed questionnaire, which is used as a measure of asthma control of a participant. Patients were asked to recall how their asthma had been during the previous week and to respond to the symptom questions on a 7-point scale (0=no impairment, 6=maximum impairment). The questions are equally weighted and the ACQ-5 score is the mean of the 5 questions: therefore, between 0 (totally controlled) and 6 (severely uncontrolled).
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS) overall population
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 299 | 293 | 298
units on scale | -0.83 (0.055) | -0.90 (0.056) | -0.71 (0.056)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.819, ANCOVA — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.27 to 0.04], Standard Error of Mean 0.079
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.591, ANCOVA — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.35 to -0.04], Standard Error of Mean 0.079

8. Secondary Outcome: Change From Baseline to Week 52 in Pre-dose Forced Expiratory Volume in 1 Second (FEV1) in Overall Population
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline is defined as the last available FEV1 measurement taken prior to the first dose of randomized study drug.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS) in overall population
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 299 | 293 | 298
Liter | 0.144 (0.0205) | 0.108 (0.0206) | 0.068 (0.0209)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.819, ANCOVA — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = 0.076, 95% CI 2-sided [0.019 to 0.134], Standard Error of Mean 0.0292
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.591, ANCOVA — adjusted p-value; Adjusted p-values obtained from the closed testing procedure; Mean Difference (Net) = 0.040, 95% CI 2-sided [-0.017 to 0.097], Standard Error of Mean 0.0292

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are presented from first dose of study treatment until last dose of study treatment plus 7 days post treatment. Serious AEs (including the All-Cause Mortality data table) are presented from first dose of study treatment until last dose of study treatment plus 30 days post treatment, up to maximum duration of 56 weeks.
Description: Any sign or symptom that occurs during the study treatment plus 7 days post treatment for adverse events and 30 days post treatment for serious adverse events.
Groups:
- QAW039 150 mg: QAW039 150 mg
- QAW039 450 mg: QAW039 450 mg
- Placebo: Placebo
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/299 | 1/293 | 2/298
Serious Adverse Events (participants affected / at risk) | 33/299 | 30/293 | 32/298
Other Adverse Events (participants affected / at risk) | 204/299 | 193/293 | 214/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150 mg (N=299) | QAW039 450 mg (N=293) | Placebo (N=298)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 0 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Megacolon (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Bacterial diarrhoea (Infections and infestations) | 0 | 1 | 0
Chronic hepatitis C (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 2 | 1
Pneumonia (Infections and infestations) | 3 | 5 | 1
Pneumonia chlamydial (Infections and infestations) | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Thoracic spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150 mg (N=299) | QAW039 450 mg (N=293) | Placebo (N=298)
Bronchitis (Infections and infestations) | 29 | 22 | 26
Lower respiratory tract infection (Infections and infestations) | 12 | 10 | 7
Nasopharyngitis (Infections and infestations) | 43 | 37 | 49
Rhinitis (Infections and infestations) | 8 | 11 | 12
Sinusitis (Infections and infestations) | 18 | 19 | 18
Upper respiratory tract infection (Infections and infestations) | 35 | 35 | 31
Upper respiratory tract infection bacterial (Infections and infestations) | 13 | 14 | 21
Urinary tract infection (Infections and infestations) | 11 | 15 | 18
Viral upper respiratory tract infection (Infections and infestations) | 29 | 26 | 26
Blood creatinine increased (Investigations) | 13 | 11 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 16 | 11
Headache (Nervous system disorders) | 28 | 22 | 24
Asthma (Respiratory, thoracic and mediastinal disorders) | 151 | 135 | 155
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT02555683/SAP_000.pdf
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT02555683/Prot_001.pdf